CLINICAL TRIAL: NCT01739842
Title: Kudzu Effects on Brain Ethanol Levels: Proton Spectroscopy Assessment
Acronym: Kudzu MRS
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding was not received for this study.
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Scott Lukas, Director, McLean Imaging Center, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-P-001780; AA10536 (Other Grant/Funding Number: NIAAA)
Record Dates: First submitted 2012-11-13; First posted 2012-12-04 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Alcohol Consumption; Cerebral Blood Flow
Keywords: Alcohol consumption; Kudzu extract; Cerebral blood flow
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kudzu extract treatment (Active Comparator): Kudzu (2 mg) will be administered as a pretreatment 2 ½ hours before a drinking session.
  During the medication week, participants will take 2 capsules three times a day for a total dose of 3 grams of kudzu.
  Interventions: Dietary Supplement: Kudzu extract
- Placebo (Placebo Comparator): Placebo will be administered as a pretreatment 2 ½ hours before a drinking session.
  During the medication week, participants will take 2 capsules three times a day.
  Interventions: Dietary Supplement: Kudzu extract

INTERVENTIONS:
Dietary Supplement: Kudzu extract
  Other Names: Kudzu root extract (NPI-031); Puerariae lobata; Alkontrol-Herbal®

SUMMARY:
This study is designed to test whether treatment with kudzu extract will increase the rate at which alcohol enters the brain as measured by rapid proton magnetic resonance spectroscopy (1H-MRS).

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and complying with the protocol
* Good physical and mental health (normal physical exam, ECG, blood and urine chemistries, no psychopathologies)
* Body Mass Index between 18-30, inclusive
* Age 21-40 years
* Moderate alcohol drinkers (less than 20 drinks/week)
* Have a stable living situation with current postal address
* No contraindications to MR scanning (see MR scanning exclusion criteria below)

Exclusion Criteria:

* Concurrent diagnosis of Axis I disorder
* Current or past alcohol dependence; may meet criteria for alcohol abuse. Other drug dependence acceptable only if greater than 3 years.
* Current drug abuse (other than alcohol or marijuana abuse). Past drug abuse is acceptable.
* Subjects cannot be actively seeking treatment for any drug or alcohol dependence.
* Subjects cannot use marijuana more than once a week. Marijuana abuse/dependence are acceptable if the use criteria is met.
* Maintained on an antipsychotic or antidepressant medication; taking prescription medications except certain short-term anti fungal agents and some tropical creams for dermal conditions.
* Tobacco use greater than 10 cigarettes per day
* History of major head trauma resulting in cognitive impairment or history of seizure disorder
* Heavy caffeine use (greater than 500 mg on a regular, daily basis)
* For female volunteers, a positive pregnancy test

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Rate at which alcohol enters the brain | 2.5 hours after drug administration
  To determine the effects of kudzu extract treatment on the rate at which alcohol enters the brain and to determine if this is due to a change in cerebral blood flow as measured by rapid proton magnetic resonance spectroscopy (1H-MRS).

SECONDARY OUTCOMES:
Impact of alcohol and kudzu on resting state networks (RSN). | 2.5 hours after drug administration